CLINICAL TRIAL: NCT04758793
Title: Muscles in Liver Diseases
Acronym: UNIVERSE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: APHP201215
Record Dates: First submitted 2021-01-07; First posted 2021-02-17 (Actual); Last update posted 2021-02-17 (Actual); Status verified 2020-12

CONDITIONS: Patients Having a Scheduled Abdominal Surgery Procedure
MeSH Terms: interventions — Blood Specimen Collection

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- patients without liver disease, (Other): taking blood samples and biopsy of muscular wall
  Interventions: Other: blood samples; Other: biopsy of abdominal paroie
- patient with chronic liver disease without cirrhosis, (Other): taking blood samples and biopsy of muscular wall
  Interventions: Other: blood samples; Other: biopsy of abdominal paroie
- patients with compensated cirrhosis, (Other): taking blood samples and biopsy of muscular wall
  Interventions: Other: blood samples; Other: biopsy of abdominal paroie
- patient with severe cirrhosis (Other): taking blood samples and biopsy of muscular wall
  Interventions: Other: blood samples; Other: biopsy of abdominal paroie

INTERVENTIONS:
Other: blood samples — 3 citrated tubes and 3 EDTA tubes
Other: biopsy of abdominal paroie — a muscle biopsy will be performed on the incision area

SUMMARY:
Cirrhosis is the 11th leading cause of death in the world. The progression to cirrhosis occurs as a result of chronic hepatic injury, related to excessive alcohol consumption, non-alcoholic steatohepatitis, chronic viral infection. Cirrhosis is accompanied by symptoms that profoundly affect the quality of life of patients.

Sarcopenia, or decrease in muscle capacity through loss of muscle mass, is associated with liver disease. Patients with liver disease and sarcopenia have increased morbidity, and higher pre- and post-liver transplant mortality than patients without sarcopenia. The mechanism responsible for the development of sarcopenia in liver disease remains largely misunderstood, as do the mechanisms by which sarcopenia appears to promote complications of liver disease.

This study, carried out on a prospective cohort of patients with liver disease, aims at understanding the pathophysiological mechanisms involved in sarcopenia and its consequences.

DETAILED DESCRIPTION:
Cirrhosis is the 11th leading cause of death in the world. The progression to cirrhosis occurs as a result of chronic hepatic injury, related to excessive alcohol consumption, non-alcoholic steatohepatitis, and chronic viral infection. Cirrhosis is accompanied by symptoms that profoundly affect the quality of life of patients.

Sarcopenia, or decrease in muscle capacity through loss of muscle mass, is associated with liver disease. Patients with liver disease and sarcopenia have increased morbidity, and higher pre- and post-liver transplant mortality than patients without sarcopenia. The mechanism responsible for the development of sarcopenia in liver disease remains largely misunderstood, as do the mechanisms by which sarcopenia appears to promote complications of liver disease.

This study, carried out on a prospective cohort of patients with stable liver disease, aims at understanding the pathophysiological mechanisms involved in sarcopenia and its consequences.

After checking the inclusion criteria, all eligible patients treated at Beaujon Hospital (Clichy) will be invited to participate in the study. After inclusion, clinical and laboratory features (hepatic assessment) will be collected and the blood samples will be taken.

During the surgery, a muscle biopsy will be performed on the incision area. No follow-up is planned.

ELIGIBILITY:
Inclusion Criteria:

* Patients over the age of 18 having a scheduled abdominal surgery at Beaujon Hospital
* Patient affiliated to a social security scheme
* Informed patient having signed a consent to participate

Exclusion Criteria:

Primary muscle disease (myopathy, dermatopolymyositis, vasculitis with muscle involvement)

* Amyotrophic drugs: long-term corticosteroid therapy
* Immunosuppressive treatments
* Chronic inflammatory disease (example: Crohn's disease)
* Disease known to cause sarcopenia such as -but not limited to- active extrahepatic neoplasia, polycystic hepatorenal disease
* Gastrointestinal haemorrhage in the 15 days prior to inclusion
* Acute alcoholic hepatitis in the month before inclusion
* Infection during treatment
* Pregnant or breastfeeding woman
* Protected populations: people under guardianship or under guardianship
* Patient not affiliated to a social security scheme
* Patient under AME
* Patient not having signed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 260 (Estimated)
Dates: Start 2021-02-15 (Estimated); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
describe the muscle changes that occur during liver disease. | 1 month after the of inclusion
  Assessment of the histology of the muscle removed during abdominal surgery by measuring the diameter of muscle fibers
describe the muscle changes that occur during liver disease. | 1 month after the of inclusion
  Assessment of the histology of the muscle removed during abdominal surgery, by evaluating the vascularity with measurements of CD31 count and αSMA count
describe the muscle changes that occur during liver disease. | 1 month after the of inclusion
  Assessment of the histology of the muscle removed during abdominal surgery by evaluating the muscle stem cells with measurements of Pax7, MyoD and Myogenin
describe the muscle changes that occur during liver disease. | 1 month after the of inclusion
  Assessment of the histology of the muscle removed during abdominal surgery by evaluating gene expression with transcriptomics

SECONDARY OUTCOMES:
Identify circulating mediators that could be responsible for sarcopenia: released by the liver and acting on the muscle. | 1 month after the of inclusion
  Circulating concentration of mediators / cells suspected of being responsible for sarcopenia:
  * extracellular vesicles released by the liver
  * lymphocyte phenotype potentially modified by sinusoidal endothelial cells of the liver
  * protein array
Identify circulating mediators that could be responsible for complications of liver disease: released by the muscle and acting on the different organs | 1 month after the of inclusion
  Circulating concentration of mediators / cells suspected of being released by muscle and contributing to organ dysfunction in liver disease:
  * extracellular vesicles
  * myokines

IPD SHARING:
Plan to Share IPD: Undecided